CLINICAL TRIAL: NCT02659839
Title: Mortality in Cancer Patients Admitted to the Intensive Care Unit in a Resource-limited Setting: A Prospective Cohort Study
Brief Title: Mortality in Cancer Patients Admitted to the Intensive Care Unit in a Resource-limited Setting
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 101015
Record Dates: First submitted 2016-01-16; First posted 2016-01-20 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Cancer
Keywords: Cancer; Intensive care unit; Mortality
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients admitted to the ICU: Patients with cancer admitted to the ICU. No intervention will be administered.
  Interventions: Other: Cancer patients admitted to the ICU

INTERVENTIONS:
Other: Cancer patients admitted to the ICU — There will be no change in the standard ICU treatment.
  Other Names: Standard intensive care unit management.

SUMMARY:
The purpose of this study is to determine 30 day mortality in cancer patients admitted to the intensive care unit in a resource limited setting.

DETAILED DESCRIPTION:
The management of cancer patients in the intensive care unit (ICU) has changed dramatically during the last two decades. Initial experiences showed high rates of hospital mortality, reaching up to 75-85% in patients requiring life-sustaining treatments, particularly mechanical ventilation. An increasing number of clinical experiences has been reported pointing to a significant improvement in survival of these patients. However, it is not clear if this results are generalizable to settings with resource constraints. Therefore, the purpose of this study is to determine 30 day mortality in cancer patients admitted to the intensive care unit in a resource limited setting.

This study is a prospective cohort of cancer patients admitted to the ICU in which the investigators will evaluate the prognostic of cancer patients admitted for a ICU trial or treatment in ICU without limitations. This study will not consider any change in the treatment plan of the patients. The source of the data will be the clinical records of the patients during the admission and the records of the cancer unit. There will be no direct contact of the research team with the patients or their family.

ELIGIBILITY:
Inclusion Criteria:

* 18 years-old or older
* Histological diagnosis or high clinical suspicious of cancer (solid /hematological), with the exception of non-melanoma skin cancer.
* Functional classification state between 0-3, according to Eastern Cooperative Oncology Group.
* Admission to intensive care unit, because of one or more of the following criteria:

  1. Invasive or non-invasive ventilatory support due to acute respiratory failure.
  2. Use of vasopressor drugs due to hypotension defined as noradrenaline requirement higher than 0.1 microgram/Kg/min.
  3. Renal replacement therapy due to acute renal failure.

Exclusion Criteria:

* Absence of cancer recurrences in more than 5 years after diagnosis
* Functional classification state of 4, according to Eastern Cooperative Oncology Group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with histological diagnosis or high clinical suspicious of cancer, admitted to the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Mortality at 30 days | 30 days since ICU admission

SECONDARY OUTCOMES:
Mortality at 180 days | 180 days since ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Sebastián Mondaca, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Dr. Sótero del Rio, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Panay S, Ruiz C, Abarca M, Nervi B, Salazar I, Caro P, Muniz S, Briones J, Bruhn A, Mondaca S. Mortality of Adult Patients With Cancer Admitted to an Intensive Care Unit in Chile: A Prospective Cohort Study. J Glob Oncol. 2018 Dec;4:1-9. doi: 10.1200/JGO.18.00091. PMID 30582431